CLINICAL TRIAL: NCT00446017
Title: Phase 3 Study of Adrenaline and Milrinone in Patients With Myocardial Dysfunction
Brief Title: The Effects of Adrenaline and Milrinone in Patients With Myocardial Dysfunction After CABG
Acronym: AMORI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL-ANAE-101
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2007-04

CONDITIONS: Cardiac Output, Low
Keywords: coronary artery bypass grafting; inotropes; metabolism; renal failure
MeSH Terms: conditions — Cardiac Output, Low; Renal Insufficiency | interventions — Epinephrine; Milrinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: adrenaline
Drug: milrinone

SUMMARY:
Myocardial dysfunction necessitating inotropic support is a typical complication after on-pump cardiac surgery. This prospective, randomized pilot-study analyses the metabolic and renal effects of the inotropes adrenaline and milrinone in patients needing inotropic support after coronary-artery-bypass-grafting. With respect to data derived from patients with sepsis shock and results from studies using phosphodiesterase-inhibitors prophylactically, the hypothesis is tested that adrenaline may be associated with unwarranted metabolic effects (hyperlactatemia and hyperglycemia) and renal dysfunction.

DETAILED DESCRIPTION:
Following preoperative written informed consent, patients presenting with a cardiac-index (CI) < 2.2 l/min/m2 upon ICU-admission - despite adequate mean arterial (titrated with noradrenaline or sodium-nitroprusside) and filling pressures - will be randomized to 14 hour treatment with adrenaline or milrinone to achieve a CI > 3.0 l/min/m2.

A group of patients not needing inotropes will be used as controls. Hemodynamics, metabolism (plasma lactate, pyruvate, glucose, acid-base status, insulin requirements) and renal function (urinary excretion of alpha-1-microglobulin, creatinine clearance, plasma cystatin-C levels) will be determined during the treatment period and up to 48 hours after surgery (follow up period).

The study is designed as a pilot study including 20 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* cardiac index below 2.2 l/min/m2 upon intensive care unit admission despite optimized filling pressures and normalized mean arterial blood pressure (MAP) after elective coronary artery bypass grafting

Exclusion Criteria:

* intraoperative use of diuretics or hydroxyethylstarch

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-06; Primary Completion 2004-08 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Plasma lactate concentration in the immediate postoperative period

SECONDARY OUTCOMES:
Hemodynamics
Plasma pyruvate
Plasma glucose
Plasma creatinine
Urinary excretion of alpha-1-microglobulin
Plasma cystatin C

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Heringlake, MD, Principal Investigator — Department of Anesthesiology, University of Luebeck

REFERENCES:
- [Derived] Heringlake M, Wernerus M, Grunefeld J, Klaus S, Heinze H, Bechtel M, Bahlmann L, Poeling J, Schon J. The metabolic and renal effects of adrenaline and milrinone in patients with myocardial dysfunction after coronary artery bypass grafting. Crit Care. 2007;11(2):R51. doi: 10.1186/cc5904. PMID 17470271